CLINICAL TRIAL: NCT05598424
Title: Establishment of CST1 Predictive Model of Oral Glucocorticoid Therapy Sensitivity for Chronic Rhinosinusitis With Polyps
Brief Title: CST1 Predictive Model of Oral Glucocorticoid Therapy Sensitivity for Chronic Rhinosinusitis With Polyps
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TR-CST1
Record Dates: First submitted 2022-10-25; First posted 2022-10-28 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyps; Glucocorticoids
MeSH Terms: interventions — Glucocorticoids; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oral Glucocorticoids group (Experimental): Intervention Period I: nasal spray, Budesonide Nasal Spray, 64ug per Nostril, bid, for 4-week duration.
  Intervention Period II: oral glucocorticoids methylprednisolone 24mg qd, and nasal spray, Budesonide Nasal Spray 64ug per Nostril, bid, for 2-week duration.
  Interventions: Drug: Oral Glucocorticoids

INTERVENTIONS:
Drug: Oral Glucocorticoids — Oral Glucocorticoids（methylprednisolone） 24mg qd, 2-week duration
  Other Names: methylprednisolone

SUMMARY:
Topical and systemic steroids constitute the first choice in medical treatment for nasal polyps. Glucocorticoids sensitivity is significantly correlated with CST1 level in nasal secretions. The goal of this single-arm clinical trial based on a multicenter platform is to test CST1 in patients with chronic rhinosinusitis and nasal polyps before and after oral glucocorticoid therapy. Endoscopic polyp score, Total Nasal Symptom Score(TNSS), SNOT-22 score and other biomarkers are also evaluated before and after the treatment. Researchers will develop a CST1 predictive model of oral glucocorticoid therapy for Chronic Rhinosinusitis with Polyps.

ELIGIBILITY:
Inclusion Criteria:

1. All meet the diagnostic criteria of CRSwNP in EPOS2020 (Age 18-70 years old);
2. Investigator-assessed endoscopic bilateral Nasal Polyp Size Score (NPSS) was greater than or equal to 4 (minimum score of 2 per nasal cavity);

Exclusion Criteria:

1. Oral glucocorticoid contraindications, such as diabetes, femoral head necrosis, gastric ulcer, etc.
2. Medication history of oral glucocorticoids or immunomodulator within 1 months before enrollment, antibiotics within 2 weeks;
3. fungal sinusitis, allergic fungal sinusitis (AFRS), cystic fibrosis, primary ciliary dyskinesia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-11-22 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
The change in endoscopic polyp score | Baseline, week 4, week 6
  Bilateral polyp volume size described using the Nasal Polyp Size Score (NPSS) score. (0 - 4 points per side: 0 = no polyp; 1 = small polyp in the middle meatus, not reaching the inferior border of the middle turbinate; 2 = small polyp in the middle meatus, reaching the inferior border of the middle turbinate; 3 = large polyp protruding from the middle meatus, not reaching the inferior border of the inferior turbinate; 4 = large polyp that almost causes most or complete obstruction of the nasal cavity.)

SECONDARY OUTCOMES:
The change in Total Nasal Symptom Score | Baseline, week 4, week 6
  Total Nasal Symptom Score was are graded on a 3-point scale. (0= no symptoms; 1= mild symptoms; 2= moderate symptoms; 3= severe symptoms).
The change in SNOT-22 score | Baseline, week 4, week 6
  The 22-item Sino-nasal outcome test (SNOT-22) was used to evaluate the changes in symptoms of patients.
  According to the severity of symptoms caused by RCRS, each item was divided into 6 levels: no distress (0 points), mild distress (1 point), mild distress (2 points) ), moderate distress (3 points), severe distress (4 points), very severe distress (5 points). The higher the score, the more severe the symptoms, and the final total score of the item is counted.
The change in asthma ACQ Score | Baseline, week 4, week 6
  For patients with asthma, we assessed the change of asthma symptoms through the Asthma Control Questionnaire(ACQ). Each question was scored on a scale of 0 to 6 according to the severity. The result score of each item was averaged. A score of <0.75 indicated that the asthma had been completely controlled; a score of 0.75-1.5 indicates well-controlled asthma; a score of >1.5 indicates that asthma is not controlled.
The change of CST1 | Baseline, week 4, week 6
  The change of Cystatin 1
The change of biomarker | Baseline, week 4, week 6
  Changes in expression levels of biomarker in nasal brush exfoliated cells, nasal secretions and nasal microbes.
The change in AE / SAE recording | Baseline, week 4, week 6
  Any adverse event
The change of inflammatory cell | week 4, week 6
  The change of inflammatory cell in nasal polyps
The change of serum cortisol | Baseline, week 4, week 6
  The change of serum cortisol level

CONTACTS AND LOCATIONS:
Overall Officials: Luo Zhang, Study Chair — Beijing Tongren Hospital
Locations (1):
- Beijing Tongren Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No